CLINICAL TRIAL: NCT07201558
Title: An Open-label, Phase I Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Surovatamig Following Single-ascending Dose and Step-up Dose Administration to Adult Participants With Rheumatoid Arthritis or Systemic Lupus Erythematosus
Brief Title: Study Evaluating Safety, Tolerability, PK/PD of Surovatamig in Adult RA or SLE Participants
Acronym: ASSURO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D740AC00001; 2025-522273-10-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-09-30; First posted 2025-10-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus
Keywords: adult participants; rheumatoid arthritis; systemic lupus erythematosus; surovatamig
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: This is an open-label study consisting of up to 3 parts: SAD (Part 1), sSUD (Part 2), and optional dSUD (Part 3). Depending on the assigned study part, participants will either receive surovatamig once (Part 1), twice (Part 2), or three times (Part 3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Surovatamig (Experimental): Participants will receive Surovatamig subcutaneously in one of three dosing regimens: once (Part 1), twice (Part 2), or three times (Part 3), depending on the study part.
  Interventions: Biological: Surovatamig

INTERVENTIONS:
Biological: Surovatamig — Surovatamig is a bispecific T-cell engager administered subcutaneously. This is an open-label, dose-escalation study evaluating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of Surovatamig in adult participants with rheumatoid arthritis (RA) or systemic lupus erythematosus (SLE). The study consists of up to three parts:
  Part 1 (SAD): Single ascending dose - participants receive one dose of Surovatamig.
  Part 2 (sSUD): Single step-up dosing - participants receive two doses. Part 3 (dSUD): Double step-up dosing - participants receive three doses. Participants are assigned to a study part based on protocol-defined criteria. The study includes follow-up for a minimum of 179 days post-first dose, with extended monitoring up to 12 months for certain participants.

SUMMARY:
This open-label, Phase I study will assess the safety and tolerability of surovatamig and characterise its PK and PD following subcutaneous administration to participants with RA or SLE.

DETAILED DESCRIPTION:
This is an open-label, Phase I, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of surovatamig administered subcutaneously in adult participants aged 18 to 65 years with rheumatoid arthritis or systemic lupus erythematosus. The study includes single-ascending and step-up dosing cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 (or the legal age of consent in the jurisdiction in which the study is taking place) to 65 years of age, inclusive, at the time of signing the informed consent.
2. For RA participants, only:

1. Diagnosis of RA as defined by the 2010 EULAR/ACR classification criteria 2. Positive for ≥ 1 disease-specific autoantibody performed by the central laboratory at screening. (a) RF (b) ACPA 3. Moderate or severe disease activity defined as ≥ 4 tender joints and ≥ 4 swollen joints (not including distal interphalangeal joints) 4. Intolerance to or inadequate response following approximately 3 month's treatment or longer to ≥2 b/tsDMARDs (with different mechanisms of action) after failing csDMARD therapy (unless csDMARD therapy is contraindicated). There is no minimum duration for taking a treatment in cases of intolerance.

5. Background standard of care is not a requirement for participation, however, the following therapies are permitted and may be continued during the study (alone or in combination): (a) Oral prednisone (or equivalent). Dose must be stable and ≤ 10mg a day for ≥ 2 weeks prior to Day 1. (b) Oral anti-malarial (e.g. hydroxychloroquine ≤ 400 mg a day). Dose must be stable for ≥ 4 weeks prior to Day 1. (c) Treatment with one of the following csDMARDs for ≥ 3 months and at a stable dose for ≥ 4 weeks prior to Day 1. (i) Methotrexate ≤ 25 mg per week, without change of route of administration for 8 weeks prior to Day 1 (ii) Sulfasalazine ≤ 3g/day (iii) Leflunomide ≤ 20 mg/day 3. For SLE participants, only:

1. Diagnosis of SLE as defined by the 2019 EULAR/ACR classification criteria
2. Positive for ≥ 1 disease-specific autoantibody performed by the central laboratory at screening. If autoantibodies are negative at screening, documented history of test results may be used. (a) ANA immunofluorescent assay test (titer ≥ 1:80) (a) Anti-dsDNA (b) Anti-Sm.
3. Moderate or severe disease activity defined as clinical SLEDAI-2K > 4
4. Intolerance to or inadequate response following approximately 3 months treatment or longer ≥ 3 SoC (includes: corticosteroids, anti-malarial drugs, calcineurin inhibitor, methotrexate, azathioprine, leflunomide, mycophenolic acid or its derivatives, cyclophosphamide, belimumab, anifrolumab, or B-cell depleting monoclonal antibodies). There is no minimum duration for taking a treatment in cases of intolerance.
5. Background standard of care is not a requirement for participation, however, the following therapies are permitted and may be continued during the study (alone or in combination): (a) Oral prednisone (or equivalent. Dose must be stable and ≤ 20mg a day for ≥ 2 weeks prior to Day 1. (b) Oral anti-malarial (eg, hydroxychloroquine ≤ 400 mg a day). Dose must be stable for ≥ 4 weeks prior to Day 1. (c) Treatment with one of the following immunosuppressive treatments. for ≥ 3 months and at a stable dose for ≥ 4 weeks prior to Day 1. (i) Methotrexate ≤ 25 mg/week, without change of route of administration for 8 weeks prior to Day 1 (ii) Mycophenolate mofetil or equivalent ≤ 2 g/day (dose must be ≤ 2 g/day for 3 months prior to Day 1) (iii) Azathioprine ≤ 200 mg/day (iv) Leflunomide ≤ 20 mg/day (v) Tacrolimus ≤ 0.1 mg/kg/day with maximum dose of 5 mg/day (vi) Cyclosporin ≤ 3 mg/kg/day with maximum dose of 200 mg/day

4. Blood B cells ≥ 50 cells/μL at screening. 5. IgG levels ≥ 6 g/L at screening.

Exclusion Criteria:

1. Any complications of disease under study that are judged by the Investigator to be life or organ threatening or to require treatments which are not permitted in the protocol, including but not limited to: (a) Active severe SLE-driven renal disease. (b) Severe lung or cardiac involvement. (c) History of, or current diagnosis of, catastrophic or severe APS (eg, diagnosis of an arterial or central/pulmonary venous clot) within 1 year prior to signing the ICF. Participants with clinically evident APS which is adequately controlled by anticoagulants or aspirin for at least 12 weeks can be recruited into the study. (d) Rapidly progressive and/or severe ILD or ILD that requires oxygen supplementation/therapy (of any type). (e) Felty's syndrome
2. History of HLH/MAS.
3. For RA participants, only:

1. Juvenile idiopathic arthritis or idiopathic arthritis diagnosed before the age of 16.

2. Axial spondylarthritis or any other disease associated with inflammatory arthritis 4. For SLE participants, only: History of active, severe or unstable neuropsychiatric SLE including, but not limited to: aseptic meningitis; cerebral vasculitis; myelopathy; demyelination syndromes (ascending, transverse, acute inflammatory demyelinating polyradiculopathy); acute confusional state; impaired level of consciousness; psychosis; acute stroke or stroke syndrome; cranial neuropathy; status epilepticus; cerebral ataxia, and mononeuritis multiplex.

5. Other active or prior documented severe, complex, autoimmune or inflammatory disorders. Exceptions to this exclusion criteria include: (a) Vitiligo or alopecia (b) Hypothyroidism stable on hormone replacement (c) Controlled type I diabetes mellitus on insulin (d) Any chronic skin condition that does not require systemic therapy (e) Celiac disease, controlled by diet alone (f) Sjögren's syndrome 6. Significant CNS co-morbidity (eg, Parkinson's, stroke, CNS vasculitis, severe brain injury, dementia, neurodegenerative diseases, cerebellar disease, epilepsy/seizure disorders, PML, severe uncontrolled mental illness, psychosis, CNS involvement of autoimmune diseases).

7. Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection.

8. Exclusion Criteria Related to Infection:

1. Any clinical suspicion or diagnosis of active infection at screening.
2. Opportunistic infection that meets criteria to be an SAE within 3 years.
3. Clinically significant chronic infection (for example osteomyelitis, bronchiectasis) with treatment completed less than 2 months prior to signing the ICF (except for chronic nail infections which are not exclusionary)
4. Any infection requiring hospitalisation or treatment with IV anti-infectives with treatment completed less than 4 weeks prior to signing the ICF.
5. Any infection requiring oral anti-infectives within 2 weeks prior to signing the ICF.
6. History of recurrent infection requiring hospitalisation or IV antibiotics (eg, 3 or more of the same type of infection, including systemic fungal infections, over the previous 52 weeks).

9. Participant with current or previous active or latent TB. 10. Participant with human immunodeficiency virus infection (confirmed by central laboratory at screening) 11. Participant with active EBV or CMV, assessed clinically. 12. Participant with evidence of chronic or active hepatitis B defined as HBsAg positive or HBcAB positive (tested at screening visit).

13. Participant with evidence of chronic or active Hepatitis C, meeting any of the criteria below: (a) HCV RNA positive or detectible at screening (b) HCV antibody positive at screening (apart from those with negative HCV RNA >12 weeks after completion of curative antiviral treatment for HCV or those with sustained negative HCV RNA 12 weeks apart following resolution of HCV infection if not treated).

14. Participant positive with COVID-19 PCR at screening. If patients test positive at screening or Day 1 but meet other eligibility criteria, they may be re-tested after ≥ 2 weeks. If this falls within the screening window, then they do not require re-screening.

15. Receipt of any of the following treatments or interventions ever: (a) TCEs (b) Bone marrow transplant (c) Stem cell transplant (d) Total lymphoid irradiation (e) CAR-T cell therapy (f) Alemtuzumab 16. For females only - currently pregnant (confirmed with positive pregnancy test), planning to become pregnant within the study period, or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-06-27 (Estimated); Study Completion 2028-06-27 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of surovatamig: Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs) | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs)
Safety evaluation of surovatamig: Frequency of dose limiting toxicities (DLTs). | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with DLTs (dose-limiting toxicities) as defined in the study protocol
Safety of surovatamig: Incidence of AEs/SAEs leading to discontinuation of surovatamig | Day 1 to end of the study (up to 52 weeks)
  Number of participants with AEs/SAEs leading to discontinuation of surovatamig
Tolerability of surovatamig: Incidence of treatment-related vital signs abnormalities | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with treatment-related vital signs abnormalities
Tolerability of surovatamig: Incidence of treatment-related clinical laboratory abnormalities | Day 1 to end of the study (up to 52 weeks)
  Number of participants with treatment-related clinical laboratory abnormalities
Tolerability of surovatamig: Number of participants with abnormal ECG | From baseline through Day 180.
  Number and percentage of participants with abnormal ECG.

SECONDARY OUTCOMES:
Serum Pharmacokinetics (PK) parameters of surovatamig - Cmax | From Day 1 through Day 180
  Maximum observed serum drug concentration (Cmax)
Absolute counts at Day 180 in blood CD20+ B-cells | Day 180
  Absolute counts in peripheral CD20+ B cells
Serum Pharmacokinetics (PK) parameters of surovatamig - AUC0-last | From Day 1 through Day 180
  Area under the serum concentration time curve from time zero to the time of last quantifiable analyte concentration (AUClast)
Serum Pharmacokinetics (PK) parameters of surovatamig - AUCinf | From Day 1 through Day 180
  Area under the serum concentration time curve from time zero to infinity (Part 1 only)
Serum Pharmacokinetics (PK) parameters of surovatamig - AUCtau | From Day 1 through Day 180
  Area under the serum concentration time curve over a dose interval (Parts 2 and 3 only)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (3):
  - Research Site, Birmingham, Alabama
  - Research Site, Fullerton, California
  - Research Site, Allen, Texas
- Australia (2):
  - Research Site, Birtinya
  - Research Site, Clayton
- Research Site, Antwerp, Belgium
- Research Site, Porto Alegre, Brazil
- China (2):
  - Research Site, Beijing
  - Research Site, Nanjing
- Germany (2):
  - Research Site, Bonn
  - Research Site, München
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Córdoba
- Ukraine (3):
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/